CLINICAL TRIAL: NCT01044511
Title: Prospective, Randomized Trial of the Effects on HRQoL, Cost-Utility and Reintervention Rate, of Nurse Home Visits, in Patients With SEMS Treated Malignant Disease in the Esophagus and Cardia.
Brief Title: Quality of Life With Esophageal Stent Trial
Acronym: QUEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Bau Mortensen (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Michael Bau Mortensen, MD, PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: QUEST- AFD A
Record Dates: First submitted 2010-01-04; First posted 2010-01-08 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Esophageal Cancer; Gastro-esophageal Junction Cancer
Keywords: Esophageal cancer; Cardia cancer; Health Related quality of Life; SEMS; Home visits
MeSH Terms: conditions — Esophageal Neoplasms | interventions — House Calls

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home visit (Experimental): After SEMS placement, 2 home visits and a phonecall are made by a specialist nurse
  Interventions: Behavioral: Home visits
- Standard (Active Comparator): Standard contact via Hotline and traditional referring methods
  Interventions: Behavioral: standard

INTERVENTIONS:
Behavioral: Home visits — home visits by specialist nurse 2 times and 1 phonecall
  Other Names: Home visit,; pro active nurse care
  Arms: Home visit
Behavioral: standard — hotline
  Other Names: Phone Hotline; After hours phone line
  Arms: Standard

SUMMARY:
The aim of this study is to compare, specialist nurse home visits in patients with inoperable cancer in the esophagus or cardia, who are palliated with Self Expanding Metal Stent, to standard patient contact with regards to quality of life, number and character of reinterventions and cost-effectiveness.

DETAILED DESCRIPTION:
The aim of this study is to compare, specialist nurse home visits in patients with inoperable cancer in the esophagus or gastro-esophageal junction (cardia), who are palliated with Self Expanding Metal Stent, to standard patient contact with regards to quality of life, number and character of reinterventions and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Malignant obstruction of esophagus or cardia treated with SEMS due to non-operable disease.

Exclusion Criteria:

* Mentally unable to fill out questionaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
HRQoL, EORTC C-30, EOS-18 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Mortensen, MD,PhD, Study Director — Afd A, OUH
Locations (1):
- Afd A, OUH, Odense, Fyn, Denmark